CLINICAL TRIAL: NCT02140866
Title: Hand Exercises for Women With Rheumatoid Arthritis and Impaired ADL Ability: an Exploratory Randomized Controlled Trial
Brief Title: Hand Exercises for Women With Rheumatoid Arthritis and Impaired ADL Ability: an Exploratory Trial
Acronym: RAHExercise
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Parker Research Institute (Other)
Collaborators: Oak Foundation (Other); Aase and Ejnar Danielsens Foundation (Other); Danish Physiotherapy Foundation (Unknown); The Danish Rheumatism Association (Other); Danish Association of Occupational Therapist (Other)
Responsible Party: Principal Investigator, Eva Ejlersen Wæhrens, Senior researcher, PhD, Parker Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 109
Record Dates: First submitted 2014-05-02; First posted 2014-05-16 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2017-09

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hand Exercise (Experimental): The intervention group will receive an exercise program for the hand/arm in combination with a compensatory intervention program (CIP).
  Interventions: Other: Hand Exercise
- Compensatory Intervention Program (CIP) (Active Comparator): The control group will receive the Compensatory Intervention Program (CIP) only.
  Interventions: Other: Compensatory Intervention Program (CIP)

INTERVENTIONS:
Other: Hand Exercise
  Arms: Hand Exercise
Other: Compensatory Intervention Program (CIP)
  Arms: Compensatory Intervention Program (CIP)

SUMMARY:
The study examines whether hand exercise therapy as an add on to a compensatory intervention program focused on joint protection, assistive devices and alternative methods of doing will improve the performance of ADL tasks requiring hand function in patients with rheumatoid arthritis (RA).

ELIGIBILITY:
Inclusion Criteria:

* Female sex.
* Age ≥ 18.
* Diagnosis of rheumatoid arthritis (2).
* Involvement of the hands, due to minimum one tender wrist, metacarpophalangeal (MCP) or proximal interphalangeal (PIP) joint in one of the hands.
* Be on stable medication for at least 3 months prior to participation.
* Self-reported decreased ability to perform personal and instrumental ADL tasks involving the hands.

Exclusion Criteria:

* Significant osteoarthritis of the hand assessed at the initial examination by the rheumatologist
* Hand surgery within 6 months of study participation
* Other pain condition involving muscles and/or joints, e.g. fibromyalgia.
* Prednisolon therapy, change in dose of biological agent or start of treatment with a new biological agent within the last 3 month before study start.
* Inability to understand the information or to speak Danish
* Any other condition that in the opinion of the investigator or accessing rheumatologist puts an otherwise eligible participant at increased risk by participation or otherwise make the person unfit for participation.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
The Assessment of Motor and Process Skills (AMPS) - the motor skill scale | within 2 weeks post intervention

SECONDARY OUTCOMES:
The Assessment of Motor and Process Skills(AMPS) - the process skill scale | within 2 weeks post intervention
The Activities of Daily Living Questionnaire (ADL-Q) | within 2 weeks post intervention
Health Assessment Questionnaire (HAQ) | within 2 weeks post intervention
Overall disease activity (DAS-28) | within 2 weeks post intervention
Grip strength | within 2 weeks post intervention

OTHER OUTCOMES:
Ultrasound Doppler | within 2 weeks post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Eva E Wæhrens, PhD, Principal Investigator — The Parker Research Institute
Locations (1):
- Copenhagen University Hospital, Frederiksberg, Frederiksberg, Denmark

REFERENCES:
- [Derived] Ellegaard K, von Bulow C, Ropke A, Bartholdy C, Hansen IS, Rifbjerg-Madsen S, Henriksen M, Waehrens EE. Hand exercise for women with rheumatoid arthritis and decreased hand function: an exploratory randomized controlled trial. Arthritis Res Ther. 2019 Jun 26;21(1):158. doi: 10.1186/s13075-019-1924-9. PMID 31242937